CLINICAL TRIAL: NCT02281864
Title: Interventions to Help Smoking Parents of Inpatients Reduce Exposure (INSPIRE)
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-0105.cc; R01CA181207-01A1 (NIH)
Record Dates: First submitted 2014-10-16; First posted 2014-11-04 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Tobacco Use Cessation; Second Hand Tobacco Smoke
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group: Quitline (Other): Quitline referral. If the family is randomized to the control group, the research team will give the parent a brochure for the QuitLine
  Interventions: Other: Control Group: Quitline
- Intervention Group (Experimental): Smoking Cessation Intervention Bundle. The Investigator has developed an intervention that bundles the best evidence for tobacco dependence treatment, including the USPHS guidelines, and evidence from parent-specific interventions, to create a sustainable, transferrable intervention specific to using the inpatient stay to help parents quit smoking and reduce their children's exposure. The intervention bundle includes screening for exposure, assessing readiness to quit, providing at least one brief motivational interviewing session in the hospital, dispensing nicotine replacement therapy if appropriate, providing a smoking cessation/reduction starter kit and arranging for follow up after the child is discharged.
  Interventions: Behavioral: Smoking Cessation Intervention Bundle

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention Bundle — Receipt of the smoke cessation/reduction intervention bundle followed by referral to the Quitline.
  Arms: Intervention Group
Other: Control Group: Quitline — Referral to the Quitline
  Arms: Control Group: Quitline

SUMMARY:
Children who are hospitalized are especially vulnerable to the effects of tobacco use and dependence among their caregivers, and they are more likely to be exposed than children who are not hospitalized. Hospitalization is an important teachable moment for health care providers to intervene with tobacco dependent parents, and help them reduce their child's exposure, potentially improving outcomes after hospitalization, and their future health. Understanding the best way to approach and intervene with these families will provide the investigator with the necessary information to create a sustainable intervention that can be disseminated to hospitals across the country that provide pediatric care, and to ultimately make a significant improvement in the health of children.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) to determine whether the proposed bundled intervention is superior to usual care in the pediatric inpatient setting can decrease children's secondhand smoke exposure, and encourage their parents to make smoke-free home rules and quit smoking, as measured by a validated survey and biomarkers.

We have developed an intervention that bundles the best evidence for tobacco dependence treatment, including the United States Public Health Service (USPHS) guidelines, and evidence from parent-specific interventions, to create a sustainable, transferrable intervention specific to using the inpatient stay to help parents quit smoking and reduce their children's exposure. The intervention bundle includes screening for exposure, assessing readiness to quit, providing at least one brief motivational interviewing session in the hospital, dispensing nicotine replacement therapy if appropriate, providing a smoking cessation/reduction starter kit and arranging for follow up after the child is discharged.

INSPIRE specific aims:

Aim 1: To assess the efficacy of the intervention in increasing parent report of having smoke-free homes and cars 6 and 12 months after hospitalization

Aim 2: To demonstrate whether children whose parents receive the intervention bundle have greater decreases in cotinine levels 6 and 12 months post-hospitalization

Aim 3: To assess the efficacy of the intervention in increasing parent quit rates 6 and 12 months after hospitalization

Aim 4 (Exploratory): To use implementation process measures from the RE-AIM framework to assess the extent that our intervention results in hospital-wide systems change, including automatic screening for tobacco smoke exposure and delivery of tobacco control services.

ELIGIBILITY:
Inclusion Criteria:

* Families admitted to the inpatient units of Children's Hospital Colorado
* Families with children <17 years of age
* Families with at least one custodial parent smoker

Exclusion Criteria:

* Admitted in the hospital < 24 hours
* Families with children in foster care
* Families with unclear custody of the child (i.e. children admitted with non-accidental trauma)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-12-10 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Demonstrate whether children whose parents receive the intervention bundle have greater decreases in cotinine levels | 12 months after patient hospitalization
  Measured by child urine cotinine levels

SECONDARY OUTCOMES:
Increased parent report of having smoke free homes and cars | 12 months after patient hospitalization
  Measured by questionnaire
Increased parent quit rates | 12 months after patient hospitalization
  Measured by questionnaire and parent urine cotinine levels
Child exposure prevalence | 12 months after patient hospitalization
  Measured by questionnaire
Child sick visits | 12 months after patient hospitalization
  Measured by data abstraction from medical record and data obtained from child's pediatrician

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Wilson, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Holstein JA, O'Hara K, Moss A, Lowary M, Kerby G, Hovell M, Klein JD, Winickoff JP, Wilson K. Barriers and Motivators for Smoking Cessation Among Caregivers of Inpatient Pediatric Patients. Hosp Pediatr. 2022 Feb 1;12(2):220-228. doi: 10.1542/hpeds.2021-005984. PMID 35083490
- [Derived] Wilson KM, Torok MR, Wei B, Wang L, Lowary M, Blount BC. Marijuana and Tobacco Coexposure in Hospitalized Children. Pediatrics. 2018 Dec;142(6):e20180820. doi: 10.1542/peds.2018-0820. PMID 30455340